CLINICAL TRIAL: NCT02884778
Title: Evaluation of the Last Version of the PMD200TM and Its NoL Index in Patients Undergoing Laparotomies With Intraoperative Epidural Analgesia
Brief Title: Observational Evaluation of the Last Version of the PMD200TM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: Medasense Biometrics Ltd (Other)
Responsible Party: Principal Investigator, Philippe Richebé, MD, PhD, Full Professor, Director of Research of the Department of Anesthesiology, Maisonneuve-Rosemont Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15074
Record Dates: First submitted 2016-07-27; First posted 2016-08-31 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Pain Monitor During Anesthesia
Keywords: pain; monitoring; anesthesia
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NoL index in response to stimulation (Experimental): There is only one arm in this study. The "intervention" is not a drug, but it is the stimulus applied to the patient such as intubation and a standardized electrical stimulus applied on the forearm of the anesthetized patient. There are several stimuli that are the so-called "interventions" and the NoL index and the classical vital signs (heart rate, mean blood pressure, BISspectral index) are registered in response to these stimuli in an observational manner.
  Interventions: Diagnostic Test: Detection of pain after nociceptive stimulus

INTERVENTIONS:
Diagnostic Test: Detection of pain after nociceptive stimulus — We will evaluate the changes of the NoL index absolute values after different types of stimulations such as intubation and electrical tetanic stimulation of the forearm (applied with the standard muscle relaxation monitor) in a patient under general anesthesia + epidural anesthesia for abdominal surgery

SUMMARY:
Title: Evaluation of the last version of the PMD200TM and its NoL index in patients undergoing laparotomies with intraoperative epidural analgesia Objectives: Measure NoL Index changes after a standardized nociceptive electrical stimulus at various intravenous remifentanil infusion rates (0.005, 0.05, 0.1 mcg/kg/min) and also after clinical stimuli such as intubation.

Study Design: Prospective observational study Subject Population: Adults scheduled to undergo elective abdominal surgery with laparotomy under general anesthesia and epidural analgesia Sample Size: 30 patients Study Duration: Starts April 2016 - Ends November 2016 Study Center: Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada Adverse Events: None expected

DETAILED DESCRIPTION:
The motivation behind the actual observational proposed study is to validate the ability of the new PMD-200TM system to accurately detect a nociceptive stimulus that occur during anesthesia (e.g. laryngoscopy for tracheal intubation, standardized electrical stimulations). The NoL index will also be recorded during period of time without any stimulation and called baseline values of NoL under standard anesthesia.

The PMD100TM was an early prototype of the pain monitor device developed by Medasense Biometrics Ltd (Ramat Yishai, Israel), which was used in our center in Montreal in a recently completed clinical trial. This device is based on a software that was integrated into a computer to analyze the different criteria with a multi-parametric index named NoL which estimates the nociception level during general anesthesia and incorporates heart rate, heart rate variability (0.15-0.4 Hz band power), plethysmograph wave amplitude, skin conductance level, number of skin conductance fluctuations (NSCF), and their time derivatives, using a non-linear regression technique. The rationale for the use of skin conductance and NSCF is that the presence of a physical stressor leads to a sympathetic-mediated filling of the palmar sweat glands, thus changing the ion concentration and the skin conductance. It has been shown to correlate with clinical stress score during intubation and to be less reactive to a tetanic stimulation when remifentanil was perfused. With the Medasense device PMD100TM, these five variables are obtained through a single non-invasive finger probe connecting the finger of the patient to the computer. Only signals from the patient are recorded. No signal is sent to the patient by the PMD100TM. The NoL Index obtained and displayed on the Medasense PMD200™ device is a single number from 0 to 100, with a lower score proposed to represent less painful stimulation.

The PMD-200TM system is an advanced configuration product in the final stages of development, with the introduction of several enhancements related to the Hardware (HW) and the Software (SW) platform:

1. Enhanced finger probe - which include 4 new sensors (slightly different from the sensors used in PMD-100 and more efficient in terms of quality of signals)
2. Improvement in the signal acquisition board - a HW module which converts the analog signals from all sensors to digital data
3. All in one system - enables integrated viewing of the recorded signals and NoL index through a touch based user interface (the previous interface for the PMD100 was on a computer screen)
4. A new Graphic user interface for the user The purpose of this new prospective observational study with the finalized PMD200TM device is to evaluate the responses of a multi-parameter index (the Nociception Level [NoL] Index) when patients under combined general anesthesia/epidural anesthesia for laparotomies are subjected to standard painful stimuli (laryngoscopy for intubation). Also during surgery, standardized electrical stimulations over the ulnar nerve (70 mA, 100 Hz for 30 seconds) at different doses of remifentanil steady state infusion (0.005 mcg/kg/min; 0.05 mcg/kg/min; 0.1 mcg/kg/min) will be performed as we did in our previous study at HMR after Scientific and Ethic Committee approval in 2015.

Studying the effect of different doses of infused remifentanil on the new and finalized version of the NoL Index from the PMD200TM device in patients subjected to a standardized painful stimulus under general anaesthesia would help validating this final version and to compare results to the prototype used in our center in a previous study.

Primary Aim: Establish a correlation between the NoL Index changes and the infused dose of remifentanil at the time the stimulation was applied. It is expected to see a strong correlation meaning that when the remifentanil infusion is high, the NoL response to the standardized electrical stimulation might be low.

Secondary Aims: NoL changes at different times of the surgery. Heart rate and blood Pressure and BISpectral index changes after clinical stimulus such as intubation, incision, and standardized electrical stimulations at different concentrations/infusions of remifentanil (0.005, 0.05, 0.1 msg/kg/min). Measure the sensitivity and specificity of the study criteria (NoL, BIS, Heart Rate and Mean Blood Pressure) in detecting a painful stimulus such as intubation and electrical stimulus at remifentanil 0.005mcg/kg/min if infusion.

Also, at the end of the surgery, we will still record the NoL index from the PMD200TM device. And we will also record the first pain score when the patient is extubated in PACU. This will be done in an observational manner. We will evaluate whether the last NoL index recorded under general anesthesia at the end of the surgical procedure (last stiches) with patient still under controlled ventilation does correlate with the first pain scores in PACU.

ELIGIBILITY:
Inclusion Criteria:

* ASA status I, II or III
* Age 18 years or older
* Elective abdominal surgery with median laparotomy under general anesthesia and epidural analgesia.

Exclusion Criteria:

* Coronary artery disease
* Serious cardiac arrhythmias (including atrial fibrillation)
* Patient refusal
* History of substance abuse
* Chronic use of psychotropic and/or opioid drugs
* Use of drugs that act on the autonomic nervous system (including β-blockers)
* History of psychiatric diseases or psychological problems
* Contraindications to epidural analgesia
* Allergy to remifentanil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Correlation between NoL index absolute values after electrical stimulus and the doses of remifentanil infused at the time of the stimulation. | Day of surgery during anesthesia
  Measure NoL Index peak value (in fact we will take an average of 7 values: the peak value and 3 values before and 3 values after the peak, time between values = 5sec) after a nociceptive electrical stimulus and evaluate the spearman correlation between NoL Values after stimulus and remifentanil doses. It is expected to see that when we increase the doses of remifentanil infusion we see a decrease in the NoL index response to the painful standardized electrical stimulus.

SECONDARY OUTCOMES:
NoL index peak absolute value after painful stimulus: intubation, electrical stimulations, no pain period, end of surgery | Day of surgery during anesthesia
  Measure NoL Index absolute peak value (in fact we will take an average of 7 values: the peak value and 3 values before and 3 values after the peak, time between values = 5sec) and delta NoL after a nociceptive stimulus such as surgical incision and standardized electrical stimulus
Heart Rate peak absolute value after painful stimulus: intubation and electrical stimulations, no pain period, end of surgery | Day of surgery during anesthesia
  Measure heart rate absolute peak value (in fact we will take an average of 7 values: the peak value and 3 values before and 3 values after the peak, time between values = 5sec) and delta heart rate after a nociceptive stimulus such as intubation and standardized electrical stimulus
Mean Arterial Blood Pressure (MABP) peak absolute value after painful stimulus: intubation and electrical stimulations, no pain period, end of surgery | Day of surgery during anesthesia
  Measure MABP absolute peak value (in fact we will take an average of 7 values: the peak value and 3 values before and 3 values after the peak, time between values = 5sec) and delta heart rate after a nociceptive stimulus such as intubation and standardized electrical stimulus
BISpectral index peak absolute value after painful stimulus: intubation and electrical stimulations, no pain period, end of surgery | Day of surgery during anesthesia
  Measure BIS absolute peak value (in fact we will take an average of 7 values: the peak value and 3 values before and 3 values after the peak, time between values = 5sec) and delta heart rate after a nociceptive stimulus such as intubation and standardized electrical stimulus
Correlation between the NoL index values (ranging from 0 to 100) and i.v. remifentanil infusion rate at the time of the electrical stimulation | Day of surgery intraoperative during anesthesia
  Establish a correlation between the NoL Index changes and the infused dose of remifentanil at the time of the standardized electrical stimulus
Correlation between the Heart Rate values and i.v. remifentanil infusion rate at the time of the electrical stimulation | Day of surgery intraoperative during anesthesia
  Establish a correlation between the Heart rate changes and the infused dose of remifentanil at the time of the standardized electrical stimulus
Correlation between the Mean Arterial Blood Pressure (MABP) values and i.v. remifentanil infusion rate at the time of the electrical stimulation | Day of surgery intraoperative during anesthesia
  Establish a correlation between the MABP changes and the infused dose of remifentanil at the time of the standardized electrical stimulus
Correlation between the Bispectral index values and i.v. remifentanil infusion rate at the time of the electrical stimulation | Day of surgery intraoperative during anesthesia
  Establish a correlation between the BIS changes and the infused dose of remifentanil at the time of the standardized electrical stimulus
Sensitivity and specificity of NoL index, Heart Rate, Mean Blood Pressure and BIS index to detect stimulus under anesthesia during surgery | Intraoperative, day of surgery
  Measure the sensitivity and specificity of the study criteria above cited in detecting a painful stimulus: intubation, electrical stimulation of the forearm.

OTHER OUTCOMES:
Correlation between end of surgery NoL value at the time of wound dressing and postoperative NRS pain scores (0-10) in PACU | Intraoperative day of surgery and day of surgery in PACU
  We will record in an observational manner the NoL index at the end of the surgery (end of wound dressing time). In PACU the first NRS score (0-10) is assessed.
  A correlation between end of anesthesia NoL index and the first NRS pain score in PACU will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Richebe, MD PhD, Principal Investigator — Hopital Maisonneuve Rosemont, CIUSSS de l'Est de l'Ile de Montreal, University of Montreal
Locations (1):
- Hopital Maisonneuve Rosemont, CIUSSS de l'Est de l'Ile de Montreal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Renaud-Roy E, Stockle PA, Maximos S, Brulotte V, Sideris L, Dube P, Drolet P, Tanoubi I, Issa R, Verdonck O, Fortier LP, Richebe P. Correlation between incremental remifentanil doses and the Nociception Level (NOL) index response after intraoperative noxious stimuli. Can J Anaesth. 2019 Sep;66(9):1049-1061. doi: 10.1007/s12630-019-01372-1. Epub 2019 Apr 17. PMID 30997633